CLINICAL TRIAL: NCT01207622
Title: Efficacy of Atomoxetine for Attention Deficit Hyperactivity Disorder (ADHD) in Adolescents and Young Adults With Substance Use Disorders (SUD)
Brief Title: Efficacy of Atomoxetine for ADHD in Adolescents and Young Adults With SUD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Timothy Wilens, MD, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-P-001823; 5K24DA016264-02 (NIH)
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Attention Deficit Hyperactivity Disorder; Substance Use Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atomoxetine (Active Comparator)
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine
  Arms: Atomoxetine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to investigate the efficacy of Atomoxetine (ATMX) in the treatments of adolescent and young adult Attention Deficit Hyperactivity Disorder (ADHD) with comorbid Substance Use Disorder (SUD). The secondary objective of the study is to determine the efficacy of ATMX in preventing SUD relapse. As previous pre-clinical work has demonstrated that ATMX has led to significant improvement in ADHD in children and lacks abuse liability, the investigators hypothesize that ATMX will be efficacious in treating ADHD in adolescents and young adults with SUD, and that ATMX will also be efficacious in preventing SUD relapse.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 15-30 years.
* Subjects with a DSM-IV diagnosis of ADHD (combined or inattentive subtype) as determined by clinical evaluation and/or ADHD module of structured diagnostic interview, completed by the study clinician.
* Subjects with a current or recent (within three months) substance use disorder (drugs or alcohol) as determined through clinical evaluation and/or ascertained through structured diagnostic interview.
* Subjects with an ADHD CGI-S of >= 4 (moderate impairment).

Exclusion Criteria:

* Pregnant or nursing females.
* Subjects with a clinically unstable medical condition that will either jeopardize patient safety or affect the scientific merit of the study, or who undergo a change in treatment during the study.
* Recent history of intravenous drug use, or subjects who have current DSM-IV criteria for abuse or dependence of cocaine, MDA, MDMA, gammahydroxybutyrate, methamphetamines, amphetamines, opioids, PCP, or benzodiazepines that in the opinion of the investigator will interfere in their ability to participate safely in the study.
* Subjects with Mental Retardation or Organic Brain Syndromes.
* Subjects who are psychotic or have a history of bipolar disorder.
* Participants who are taking any psychotropic or anti-SUD medications will be excluded from the study.
* Current DSM-IV diagnosis of major depression, depressive disorders, or anorexia as manifested by clinical interviews.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wilens, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States